CLINICAL TRIAL: NCT04762667
Title: Preoperative Planning for Reverse Shoulder Arthroplasty Using Individual Planing Strategy
Brief Title: Individual Preoperative Planning for RSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180195
Record Dates: First submitted 2021-01-28; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-01

CONDITIONS: Shoulder Osteoarthritis; Proximal Humeral Fracture; Avascular Necrosis of Humerus
Keywords: reverse shoulder arthroplasty; patient-specific instrumentation; preoperative planning
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients will undergo reverse shoulder arthroplasty with patient-specific instrumentation. (Experimental): The patients underwent preoperative planning. A 3D model was made based on CT. The optimal position of the components of the endoprosthesis has been calculated. patient-specific instrumentation were created for each scapula and humerus using 3D modeling software. Individual guides use during operation for exact position of the components of the endoprosthesis.
  Interventions: Procedure: reverse shoulder arthroplasty
- Patients will undergo conventional reverse shoulder arthroplasty. (Other): This group of patients was examined according to the standard method, Rg and CT of the shoulder joint were performed. According to the study, the sizes of the endoprosthesis were selected. Installation of the components of the endoprosthesis during the operation was carried out using standard (included in the set) guides. Orientation was performed according to the anatomical landmarks of the glenoid and the neck of the humerus, without taking into account the individual characteristics of the bones.
  Interventions: Procedure: reverse shoulder arthroplasty

INTERVENTIONS:
Procedure: reverse shoulder arthroplasty — In our work, all patients are performs MSCT of the shoulder joint. The construction of a 3D model is carried out using the obtained data. Taking into account the individual features of the bone structure of the shoulder joint, images of the pilot wire guides, fixing screws and a resection template for the humerus are created. Holes for fixing spokes for the planned structures are also calculated.
  Using a 3D printer, models of guides and a resection template are printed. During the reverse shoulder arthropalsty, instead of a standard guide, patient-specific instrumentation are used.
  In the early postoperative period, all patients are performs MSCT of the shoulder joint. The obtained data are compared with the results of MSCT of the shoulder joints of patients previously operated on using the standard technique.

SUMMARY:
Degenerative diseases and traumatic injuries of the shoulder joint, lead to dysfunction of the arm. Arthroplasty has recently become an increasingly popular operation for severe damage to the shoulder joint. In clinical practice, the most effective operation today is the reverse shoulder arthroplasty (RSA), after the installation of which the pain syndrome disappears in patients and a satisfactory range of motion in the shoulder joint resumes. With the increasing use of reverse shoulder arthroplasty and its expanding indications, surgeons today are facing tougher reconstructive challenges while still providing the patient with a good clinical outcome. The damaged joint presents a problem for the surgeon during component positioning. Implants must place the in a location and orientation that optimizes range of motion and stability while minimizing impingement. In order to address this, surgeons can look to the use of 3D imaging in order to better understand each patient's pathology.

All patients are performed computed tomography scans (CT) of the shoulder joint. Then, were reconstructed 3D model. To determine the position of the components is mounted a scapular plane was created based on 3 points on the 3D reconstructed scapula: center of the glenoid fossa, most medial point on the spinal border of the scapula, and most distal point on the inferior angle of the scapula. The investigators use a scapular plane for to determine the optimal angles of inclination of the reverse baseplate. Then the position and direction of the pilot pin is determined. The position of the fixing screws and their length are also calculated. A resection line is planned for the humerus.

Preoperative virtual templating can be used to translate the preoperative plan into the operating suite in the form of patient specific instrumentation (PSI) and intraoperative navigation. PSI to reference the local anatomy in order to place the guide pin in the desired location, version, and inclination based on the preoperative plan. After surgery, all patients undergo a CT scan of the shoulder joint. These data are compared with CT scan of patients operated on according to the standard method. The range of motion is also assessed and compared.

DETAILED DESCRIPTION:
Background: Degenerative diseases and traumatic injuries of the shoulder joint, lead to dysfunction of the arm. Arthroplasty has recently become an increasingly popular operation for severe damage to the shoulder joint. In clinical practice, the most effective operation today is the reverse shoulder arthroplasty (RSA), after the installation of which the pain syndrome disappears in patients and a satisfactory range of motion in the shoulder joint resumes. With the increasing use of reverse shoulder arthroplasty and its expanding indications, surgeons today are facing tougher reconstructive challenges while still providing the patient with a good clinical outcome. The damaged joint presents a problem for the surgeon during component positioning. Implants must place in a location and orientation that optimizes range of motion and stability while minimizing impingement. In order to address this, surgeons can look to the use of 3D imaging in order to better understand each patient's pathology.

Purpose: show the effectiveness of accurate preoperative planning and prove it using patient-specific instrumentation.

Methods: Patients aged 18 and older, male and female, are participating in our study. The established diagnosis: multifragmental fracture of the humerus head; aseptic necrosis of the humerus head; complete tears of the rotator cuff; arthrosis of the shoulder joint; rheumatoid arthritis of the shoulder joint. The study included 65 shoulders with shoulder joint pathology. The main group included 15 patients. This group of patients will undergo reverse shoulder arthroplasty with patient-specific instrumentation. Second group of patients will undergo conventional reverse shoulder arthroplasty.

In investigators work, all patients are performs MSCT of the shoulder joint, clinical assessment of the shoulder joint and assessment of neurological status.

The planning of the position of the endoprosthesis components in the main group of patients was carried out in several stages. The first stage: the position of the guide wire was calculated, taking into account the individual anatomy of the patient. The second step is to measure the angle of the pilot spoke in the axial projection. In the third stage, the planting depth is estimated. It is necessary to strive for complete adherence of the component, but at the same time, one should not forget about the preservation of the glenoid bone mass. At the fourth stage, the position of the fixing screws was calculated. Given the angle of inclination of the screws of 30 degrees, it is necessary to design the position of the screws on the 3D model so that they are as deep as possible in the bone mass. Due to this, we will obtain a reliable fixation for the glenoid base. Then we measure the length of the bone canals for the screws. The fifth stage is to calculate the direction of resection of the humeral head. For this, in a direct projection in the area of the anatomical neck, an angle of 135 degrees is built relative to the central axis of the bone.

Construction of a 3D model is carried out using the obtained data first group patients. Taking into account the individual features of the bone structure of the shoulder joint, images of the pilot wire guides, fixing screws and a resection template for the humerus are created. Holes for fixing spokes for the planned structures are also calculated.

Using a 3D printer, models of guides and a resection template are printed. During the reverse shoulder arthropalsty, instead of a standard guide, patient-specific instrumentation are used for first group patients.

In the early postoperative period, all patients are performs MSCT of the shoulder joint. The obtained data are compared with the results of MSCT of the shoulder joints of patients previously operated on using the standard technique. Functional outcomes are assessed according to the Constant-Murley Score, the University of California, Los Angeles Shoulder Assessment, and (Shoulder assessment form american shoulder and elbow surgeons, (ASES) Shoulder Outcome Score). Functional results are seen after 1, 6 and 12 months.

Planned results: in this study, we hope to prove the effectiveness of preoperative planning. The investigators expect that the precise positioning of the components using patient-specific instrumentation will increase the range of motion in the shoulder joint, reduce the complication rate, and also improve the quality of life of patients after reverse shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis: multifragmental fracture of the humerus head; aseptic necrosis of the humerus head; arthrosis of the shoulder joint.

Must be have pain and limitation of movement of the shoulder joint.

Exclusion Criteria:

massive glenoid injury. Damage to the deltoid muscle.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
MSCT after RSA. | up to 24 weeks
  postoperative MSCT data will be used for our endpoint in early postoperative period

SECONDARY OUTCOMES:
Functional outcomes are assessed according to the Constant-Murley Score | 6 months.
  assessment of the general condition, functional status of a normal or damaged shoulder joint. It consists of a section for both objective and subjective assessment, subdivided into sub-items including pain (maximum 15 points), daily activity (maximum 20 points), range of motion (maximum 40 points) and limb strength (maximum 25 points). The higher the indicator, the correspondingly better the function (minimum 0, maximum 100).
Functional outcomes are assessed according to the University of California, Los Angeles Shoulder Assessment | 6 months.
  The questionnaire includes scores for pain assessment (from 1 to 10) and function (from 1 to 10). Additionally, active anterior flexion is scored from 0 to 5 points, active flexion strength is 0-5 points, patient satisfaction is 0-5 points. Strength and range of motion are assessed by a doctor or physiotherapist, the rest of the parameters are assessed by the patient himself.
  The highest score can reach 35 points, the result above 27 points is assessed as good / excellent (satisfactory), below 27 - poor (unsatisfactory)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay A. Sukharev, Study Chair — university clinical hospital № 1I.M.Sechenov First Moscow State Medical University. Moscow, Russia
Locations (1):
- I.M. Sechenov First Moscow State Medical University (Sechenov University), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No